CLINICAL TRIAL: NCT01031940
Title: Comparison of the CMAC® Device to the Airtraq® and the Macintosh Laryngoscope in Patients With Anatomical Characteristics Predictive of Difficult Tracheal Intubation.
Brief Title: CMAC® Versus Airtraq® and Macintosh Laryngoscope in Difficult Tracheal Intubation.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Recruitment. Findings of concurrent study in low risk population not supportive of hypotheses in this study.
Sponsor: University College Hospital Galway (Other)
Responsible Party: Principal Investigator, John Laffey, Professor of Anaesthesia, University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMAC-1
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Airway; Difficult Intubation; Airway Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- macintosh (Active Comparator)
  Interventions: Device: macintosh laryngoscope
- C-MAC (Active Comparator)
  Interventions: Device: C-MAC laryngoscope
- Airtraq (Active Comparator)
  Interventions: Device: Airtraq device

INTERVENTIONS:
Device: macintosh laryngoscope — intubate with the macintosh laryngoscope
  Arms: macintosh
Device: C-MAC laryngoscope — intubate with the C-MAC laryngoscope
  Arms: C-MAC
Device: Airtraq device — intubate with the Airtraq device
  Arms: Airtraq

SUMMARY:
It is essential that anaesthetists successfully perform orotracheal intubation in scenarios in which intubation is potentially more difficult, such as where anatomical characteristics predictive of difficult intubation are present.

The CMAC® Laryngoscope is a new intubating device. It is designed to provide a view of the glottis without alignment of the oral, pharyngeal and tracheal axes.

The CMAC may be especially effective in situations where intubation of the trachea is potentially difficult.

The efficacy of this device in comparison to the traditional Macintosh laryngoscope and other novel laryngoscopes is not known.

We aim to compare its performance to that of the Macintosh laryngoscope, the gold standard device, in patients with one or more anatomical characteristics predictive of difficult intubation.

The investigators further aim to compare it to the Airtraq® device a device which has been shown to be superior to the Macintosh laryngoscope in previous trials.

The investigators primary hypothesis is that, in the hands of experienced anaesthetists, time to intubation would be shorter using the CMAC than using the Macintosh laryngoscope in patients with two or more anatomical characteristics predictive of difficult intubation.

The investigators further hypothesize that the Airtraq® will be superior the CMAC® with one or more anatomical characteristics predictive of difficult intubation.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3 patients undergoing surgical procedures requiring orotracheal intubation.
* Written informed Consent
* No relevant drug allergies
* Patients with 2 or more of the following predictors of difficult intubation:

  * Mallampatti II - IV
  * Thyromental distance < 6cm
  * Mouth opening < 3.5 cm
  * Cervical spine disease
  * Anteriorly protruding incisors
  * Presence of Caps or Crowns

Exclusion Criteria:

* Patients with history of or risk factors for gastric regurgitation
* Patients unable to consent for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Rate of successful placement of Tube in the Trachea | immediately

SECONDARY OUTCOMES:
1. Duration of Intubation attempt (successful Attempts only) a. Absolute time taken to perform successful tracheal intubation b. Number of successful intubations completed within 30 seconds | immediately
2. Tracheal Intubation attempts. a. Overall number of attempts at Intubation. b. Number of successful intubations on first attempt | immediately
3. Laryngeal View Obtained c. Cormac and Lehane Grading of Best Laryngeal View d. Change in view compared to initial assessment by independent anaesthetist. e. POGO score. | immediately

CONTACTS AND LOCATIONS:
Locations (1):
- Galway University Hospital, Galway, Galway, Ireland